CLINICAL TRIAL: NCT05640908
Title: Pelvic Fixation and Fusion During Multilevel Spinal Surgery
Acronym: PAULA
Status: Active, not recruiting | Type: Observational
Sponsor: SI-BONE, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 301106
Record Dates: First submitted 2022-11-28; First posted 2022-12-07 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Spinal Fusion; Deformity of Spine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Prospective: Participants who have scheduled spinal fusion with pelvic fixation/fusion using iFuse Bedrock Granite. These participants will be followed for 2 years.
  Interventions: Device: iFuse Bedrock Granite Implant System

INTERVENTIONS:
Device: iFuse Bedrock Granite Implant System — Surgical procedure of the spine with pelvic fixation/fusion using iFuse Bedrock Granite
  Other Names: GRANITE; Bedrock Granite

SUMMARY:
PAULA aims to collect data on the safety, performance, and effectiveness of iFuse Bedrock Granite (GRANITE) in patients who have spinal fusion surgery with pelvic fixation/ fusion.

DETAILED DESCRIPTION:
PAULA is a multicenter, open label, single-arm observational clinical study consisting of prospective and retrospective study cohorts. The goal of the study is to collect data on the safety, performance, and effectiveness of GRANITE.

ELIGIBILITY:
Inclusion Criteria:

1. ≥ 18 years of age at screening.
2. Patient is scheduled for spinal fusion with pelvic fixation/fusion using iFuse Bedrock Granite
3. Patient is willing and able to provide written informed consent

Exclusion Criteria:

1. Any known anatomic issues or permanent implants already in the pelvis that could interfere with placement of the study device(s)
2. Prominent neurologic or uncontrolled psychiatric condition that would interfere with study participation
3. Known allergy to titanium or titanium alloys
4. Current local or systemic infection that raises the risk of surgery
5. Currently pregnant or planning pregnancy in the next 2 years
6. Known or suspected active drug or alcohol abuse, including opioids
7. Patient is a prisoner or ward of the state
8. Patient is enrolled in an investigational clinical trial related to the spine

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with spinal fusion including pelvic fixation/fusion using GRANITE
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2023-06-05 (Actual); Primary Completion 2027-11 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Postoperative incidence of serious adverse events probably or definitely related to GRANITE | 2 years
Postoperative incidence of SI joint pain in subject without SI joint pain at baseline | 2 years
Postoperative incidence of L5-S1 pseudoarthrosis | 2 years
Postoperative incidence of pelvic construct failure | 2 years
  Failure is defined as:
  * Breakage of any implants placed into sacrum or ilium
  * Rod breakage in the lumbosacral region
  * Pelvic implant loosening that either causes new or worsened pain or requires surgical adjustment/revision
Postoperative incidence of device failures related to GRANITE (e.g., rod disengagement, screw pullout) | 2 years
Radiographic | 12 month and 24 months
  Bony apposition to the implant at 12 and 24 months as assessed by CT scan
Change in Quality of Life PROs | 6 month, 12 month and 24 months
  Scores on PROs at follow up timepoints compared to baseline

CONTACTS AND LOCATIONS:
Overall Officials: Robyn Capobianco, PhD, Study Director — SI-BONE, Inc.
Locations (9):
- United States (9):
  - USA Neurosurgery, Mobile, Alabama
  - University of Colorado School of Medicine, Aurora, Colorado
  - Corewell Health, Royal Oak, Michigan
  - University of Minnesota, Minneapolis, Minnesota
  - University at Buffalo, Buffalo, New York
  - Northwell Health, New York, New York
  - Pinehurst Surgical Clinic, Pinehurst, North Carolina
  - University of Texas Health, Houston, Houston, Texas
  - Texas Back Institute, Plano, Texas

IPD SHARING:
Plan to Share IPD: No